CLINICAL TRIAL: NCT04283682
Title: The Effect of Early Skin Contact Combined With Breastfeeding on Oral Feeding in Premature Infants ≤30 Weeks of Gestation
Brief Title: Intervention Facilitates Oral Feeding in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EKYY-2019-295
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Premature
Keywords: Skin Contact; bresatfeeding; premature; oral feeding
MeSH Terms: conditions — Premature Birth | interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (No Intervention): Feeding procedures follow clinical nursing practices
- intervention group (Experimental): At appropriate time to invite mothers of premature infants into the NICU for skin-to-skin and breastfeeding
  Interventions: Behavioral: Early skin-to-skin combined with breast-feeding

INTERVENTIONS:
Behavioral: Early skin-to-skin combined with breast-feeding — Premature infants in the intervention group have access to skin-to-skin once a day for 1 hour at least once no ventilation support needed. During the skin-to-skin period,the breastfeeding is encouraged for about 5-10 minutes. The whole intervention stop until the baby achieve the full oral feeding.
  Arms: intervention group

SUMMARY:
Skin-to-skin combined with breastfeeding shortened the cycle of full-oral feeding in premature infants

DETAILED DESCRIPTION:
This study is conducted at the level 3 NICU of the Children's Hospital of Fudan University, Shanghai, People's Republic of China, a tertiary medical center. Infants admitted to the NICU are all outborn infants.

The study is approved by the Ethics Committee of the Children's Hospital of Fudan University. Signed parental consent is obtained before participants'entry into the study. The RCT is conducted to evaluate the effectiveness of skin-to-skin combined with breastfeeding reduce the transition time from tube feeding to independent oral feeding.

The recruited infants are assigned to intervention group and control group.

Data are presented as means ± sds for continuous variables with normal distribution and percentages (%) for categorical variables. One-way analysis of variance and Fisher exact test is used to compare infants' baseline characteristics among the two groups. All statistical analyses are conducted using SPSS. A p value of less than 0.05 is regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≤30 weeks
* birth weight < 1500g
* age of admission <72 hours
* no congenital malformation

Exclusion Criteria:

* OI > 40
* mother has trouble in communicating

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Transition time from the initiation oral feeding to full oral feeding | During the procedure
  Transition time was defined as the days needed from introduction of oral feeding to obtain autonomous oral feeding when the nasogastric tube was removed and all the daily milk volume was taken from the bottle.

SECONDARY OUTCOMES:
Exclusive breastfeeding at discharge | During the hospitalization, an average of 2 to 3 months
  Exclusive breastfeeding at discharge is defined as through breastfeeding without bottle feeding at discharge.On the day of discharge, newborns are weighed before regular feeding and then breastfed by their mothers. After breastfeeding, the baby is weighed again and the amount of breast milk obtained by sucking the mother's breast is assessed. If the two weight subtractions are greater than or equal to the amount required for once bottle feeding, the baby is considered exclusively breastfeding at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: ling li Li, Study Chair — Wanyuan Road 399,Minhang District, Shanghai,China
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Derived] Li L, Wang L, Niu C, Liu C, Lv T, Ji F, Yu L, Yan W, Dou YL, Wang Y, Cao Y, Huang G, Hu X. Early skin contact combined with mother's breastfeeding to shorten the process of premature infants </= 30 weeks of gestation to achieve full oral feeding: the study protocol of a randomized controlled trial. Trials. 2021 Sep 17;22(1):637. doi: 10.1186/s13063-021-05605-x. PMID 34535164